CLINICAL TRIAL: NCT00590135
Title: The Effect of Statin Therapy (Atorvastatin) on the Progression of Calcific Valvular Aortic Stenosis
Brief Title: The Effect of Lipitor on Aortic Stenosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor Reducibility - primary endpoint measure not obtainable
Sponsor: The Cleveland Clinic (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 3516
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Aortic Valve Stenosis
Keywords: calcific aortic valve stenosis; echocardiography, transthoracic
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AORTIC STENOSIS PATIENTS (Experimental): Atorvastatin (Lipitor) 40mg by mouth daily is administered to patients with aortic stenosis
  Interventions: Drug: atorvastatin (Lipitor)

INTERVENTIONS:
Drug: atorvastatin (Lipitor) — atorvastatin 40 mg by mouth once daily
  Other Names: Lipitor

SUMMARY:
The purpose of this study is to find out if an approved medicine that is used to lower cholesterol called Lipitor can slow or stop progressive narrowing of the aortic heart valve in patients with a condition called aortic stenosis. Patients who have aortic stenosis who volunteer for this study will take Lipitor for 2 years and will undergo a brief exam by a physician, labwork to measure cholesterol, and a routine heart ultrasound (sound picture of the heart) at the start of the study and every 6 months, stopping at 2 years.

DETAILED DESCRIPTION:
This is a prospective, single-center study assessing the effect of atorvastatin 40 mg/day (Lipitor, Pfizer) on the progression of calcific aortic stenosis in approximately 70 patients with mild to moderate calcific AS of a tricuspid or bicuspid aortic valve. As a control population, published data on historical AS cohorts will be used, employing the accepted rate of progression of a decrease in aortic valve area of 0.1 cm²/year. Additionally, also for comparison, we will prospectively study a registry of AS patients who meet our entry criteria but are either currently already being treated with or refuse to take an HMG-CoA reductase inhibitor (referred to as the "standard care" group).

All patient visits, laboratory studies, and echocardiograms will be performed at the Cleveland Clinic Foundation in Cleveland, Ohio with the exception of the 12-week visit ALT measurement which may be done at the patient's local doctor's office and the results faxed to Imaging Research. The 12-week follow-up assessment may be completed over the phone to establish any change in patient status since baseline, study medication compliance, concomitant medication use and to ascertain whether or not the appropriate laboratory test was obtained. Over a 2-year period, assessments will be conducted at baseline, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate calcific AS of a tricuspid or bicuspid aortic valve
* Echocardiographic derived mean pressure gradient >10 mmHg and an aortic valve area of 0.9 to 1.7 cm2 by continuity equation.
* Laboratory evidence of LDL-c>70 mg/dl within 12 months prior to recruitment.

Exclusion Criteria:

* Left ventricular ejection fraction <50%
* Valvular area of 0.9 cm2 and a mean gradient >30 mmHg
* Rheumatic heart disease
* >Moderate (2+) aortic insufficiency
* Prior statin therapy to include: >10 mg of atorvastatin (Lipitor) or >20 mg of other HMG-CoA Reductase Inhibitors (statins)
* End-stage renal disease (ESRD)
* History of thoracic radiation
* Unable or unwilling to sign informed consent
* Unable to unwilling to return for follow-up
* Other clinically important renal, pulmonary, hepatic, neurological, endocrine, or hematological disorders, vasculitis, or any other situation or medical condition that, in the investigator's opinion, would make survival for the duration of the study unlikely, or would otherwise interfere with optimal participation in the study or produce a significant risk to the patient
* Severe pulmonary hypertension (>55 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2000-08 (Actual); Primary Completion 2010-04-26 (Actual); Study Completion 2010-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Griffin, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Passik CS, Ackermann DM, Pluth JR, Edwards WD. Temporal changes in the causes of aortic stenosis: a surgical pathologic study of 646 cases. Mayo Clin Proc. 1987 Feb;62(2):119-23. doi: 10.1016/s0025-6196(12)61880-1. PMID 3807436
- [Background] Walton KW, Williamson N, Johnson AG. The pathogenesis of atherosclerosis of the mitral and aortic valves. J Pathol. 1970 Jul;101(3):205-20. doi: 10.1002/path.1711010302. No abstract available. PMID 4098425
- [Background] Otto CM, Kuusisto J, Reichenbach DD, Gown AM, O'Brien KD. Characterization of the early lesion of 'degenerative' valvular aortic stenosis. Histological and immunohistochemical studies. Circulation. 1994 Aug;90(2):844-53. doi: 10.1161/01.cir.90.2.844. PMID 7519131
- [Background] Kawaguchi A, Miyatake K, Yutani C, Beppu S, Tsushima M, Yamamura T, Yamamoto A. Characteristic cardiovascular manifestation in homozygous and heterozygous familial hypercholesterolemia. Am Heart J. 1999 Mar;137(3):410-8. doi: 10.1016/s0002-8703(99)70485-0. PMID 10047619
- [Background] O'Brien KD, Reichenbach DD, Marcovina SM, Kuusisto J, Alpers CE, Otto CM. Apolipoproteins B, (a), and E accumulate in the morphologically early lesion of 'degenerative' valvular aortic stenosis. Arterioscler Thromb Vasc Biol. 1996 Apr;16(4):523-32. doi: 10.1161/01.atv.16.4.523. PMID 8624774
- [Background] Chan KL, Ghani M, Woodend K, Burwash IG. Case-controlled study to assess risk factors for aortic stenosis in congenitally bicuspid aortic valve. Am J Cardiol. 2001 Sep 15;88(6):690-3. doi: 10.1016/s0002-9149(01)01820-3. No abstract available. PMID 11564401
- [Background] Hofmann T, Kasper W, Meinertz T, Spillner G, Schlosser V, Just H. Determination of aortic valve orifice area in aortic valve stenosis by two-dimensional transesophageal echocardiography. Am J Cardiol. 1987 Feb 1;59(4):330-5. doi: 10.1016/0002-9149(87)90808-3. PMID 3812284
- [Background] Stoddard MF, Arce J, Liddell NE, Peters G, Dillon S, Kupersmith J. Two-dimensional transesophageal echocardiographic determination of aortic valve area in adults with aortic stenosis. Am Heart J. 1991 Nov;122(5):1415-22. doi: 10.1016/0002-8703(91)90585-6. PMID 1951006
- [Background] Otto CM, Pearlman AS, Gardner CL. Hemodynamic progression of aortic stenosis in adults assessed by Doppler echocardiography. J Am Coll Cardiol. 1989 Mar 1;13(3):545-50. doi: 10.1016/0735-1097(89)90590-1. PMID 2918158
- [Background] Roger VL, Tajik AJ, Bailey KR, Oh JK, Taylor CL, Seward JB. Progression of aortic stenosis in adults: new appraisal using Doppler echocardiography. Am Heart J. 1990 Feb;119(2 Pt 1):331-8. doi: 10.1016/s0002-8703(05)80024-9. PMID 2301222
- [Background] Faggiano P, Ghizzoni G, Sorgato A, Sabatini T, Simoncelli U, Gardini A, Rusconi C. Rate of progression of valvular aortic stenosis in adults. Am J Cardiol. 1992 Jul 15;70(2):229-33. doi: 10.1016/0002-9149(92)91280-h. PMID 1626512
- [Background] Peter M, Hoffmann A, Parker C, Luscher T, Burckhardt D. Progression of aortic stenosis. Role of age and concomitant coronary artery disease. Chest. 1993 Jun;103(6):1715-9. doi: 10.1378/chest.103.6.1715. PMID 8404089

RESULTS

PARTICIPANT FLOW:
Groups:
- AORTIC STENOSIS PATIENTS: Patients with mild to moderate calcific aortic stenosis will receive atorvastatin 40 mg by mouth once daily
  atorvastatin (Lipitor): atorvastatin 40 mg by mouth once daily
Period: Overall Study
Arm/Group | AORTIC STENOSIS PATIENTS
Started | 59
Completed | 0
Not Completed | 59
Not completed — Primary endpoint measure not obtainable | 59

BASELINE CHARACTERISTICS:
Arm/Group | AORTIC STENOSIS PATIENTS
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Aortic Stenosis
Description: aortic valve area as measured by transthoracic echocardiography was not obtained due to poor reproducibility
Time Frame: 2 years
Population: Population had aortic stenosis, however the primary endpoint of Aortic Valve Area was not obtainable due to poor reproducibility. As a result, the study was terminated.
Arm/Group | AORTIC STENOSIS PATIENTS
Number analyzed (Participants) | 0

2. Secondary Outcome: Rate of Change in the Aortic Valve Area Measured by Transthoracic Echocardiography Compared to That of Historical Controls
Description: Rate of change in the aortic valve area measured by transthoracic echocardiography compared to that of historical controls was not obtained. Primary outcome measurement was not obtainable, thus comparison to historic controls was not possible.
Time Frame: 2 years
Population: Primary outcome measurement was not obtainable, thus comparison to historic controls was not possible.
Arm/Group | AORTIC STENOSIS PATIENTS
Number analyzed (Participants) | 0

3. Secondary Outcome: Rate of Change in the Aortic Valve Area Measured by TEE Compared to That of Historical Controls
Description: Poor reducibility of aortic valve area measurements with transthoracic echocardiography images resulted in primary measure not being obtained. As the outcome measurement was not obtained, comparison to historical controls was not possible.
Time Frame: 2 years
Population: Poor reducibility of aortic valve area measurements with transthoracic echocardiography images resulted in primary measure not being obtained. As the outcome measurement was not obtained, comparison to historical controls was not possible.
Arm/Group | AORTIC STENOSIS PATIENTS
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Change in Aortic Valve Area as Measured by TEE Compared to Standard of Care Group
Description: Poor reducibility of aortic valve area measurements with transthoracic echocardiography images resulted in the primary outcome measure not being obtained. Thus, comparison to the stand of care group was not possible.
Time Frame: 2 years
Population: Poor reducibility of aortic valve area measurements with transthoracic echocardiography images resulted in the primary outcome measure not being obtained. Thus, comparison to the stand of care group was not possible.
Arm/Group | AORTIC STENOSIS PATIENTS
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Mean and Peak Gradients Across the Aortic Valve as Measured by TEE in the Treated Group Compared to Historical Control Group.
Description: Poor reducibility of aortic valve area measurements with transthoracic echocardiography images resulted in the primary outcome measure not being obtained. This secondary measurement was not obtained as it was deemed not relevant in the absence of the primary outcome measurement and other secondary outcome measurements.
Time Frame: 2 years
Population: Poor reducibility of aortic valve area measurements with transthoracic echocardiography images resulted in the primary outcome measure not being obtained. This secondary measurement was not obtained as it was deemed not relevant in the absence of the primary outcome measurement and other secondary outcome measurements.
Arm/Group | AORTIC STENOSIS PATIENTS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | AORTIC STENOSIS PATIENTS
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes